CLINICAL TRIAL: NCT02562417
Title: Impact of iv Dexamethasone on Reversal of Rocuronium-induced Neuromuscular Block by Sugammadex
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change of practice in the department
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 478/14
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Saline Solution; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No IV dexamethasone (Placebo Comparator): Patients will receive an equivalent volume of normal saline.
  Interventions: Drug: Normal saline
- IV dexamethasone (Experimental): Patients will receive 0.1 mg/kg of dexamethasone.
  Interventions: Drug: IV dexamethasone

INTERVENTIONS:
Drug: Normal saline
  Arms: No IV dexamethasone
Drug: IV dexamethasone
  Arms: IV dexamethasone

SUMMARY:
Sugammadex is used as a reversal drug for rocuronium- or vecuronium-induced neuromuscular block during general anaesthesia. IV dexamethasone is injected as a prophylactic measure against postoperative nausea and vomiting. Recent animal data have shown that dexamethasone may impair the reversal effect of sugammadex. The objective of this randomised controlled trial is to confirm in the clinical practice these preliminary results.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo microlaryngoscopy and ear-nose-throat endoscopic procedures

Exclusion Criteria:

* contraindication to dexamethasone administration
* contraindication to sugammadex administration
* contraindication to rocuronium administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mean recovery time for T4/T1 ratio > 90% after sugammadex administration | surgical procedure

SECONDARY OUTCOMES:
Mean recovery time for T4/T1 ratio > 80% after sugammadex administration | surgical procedure
Mean recovery time for T4/T1 ratio > 70% after sugammadex administration | surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland